CLINICAL TRIAL: NCT05422118
Title: Ascitic Fluid Calprotectin as an Accurate Diagnostic Marker for Spontaneous Bacterial Peritonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Saber Mohamed, resident doctor at clinical pathology department at faculty of medicine sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-06-07
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Active Comparator): people who have spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: ascitic fluid calprotectin
- control (Active Comparator): people who donot have spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: ascitic fluid calprotectin

INTERVENTIONS:
Diagnostic Test: ascitic fluid calprotectin — ascitic fluid calprotectin

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is an infection of the ascitic fluid in patients with liver cirrhosis and portal hypertension. There is no obvious surgical cause as perforation or intraabdominal inflammatory focus as abscess. Up to 30% of the ascitic patients will develop SBP.

SBP is attributed to immune dysfunction, bacterial translocation, circulatory dysfunction and inflammatory status. SBP is diagnosed by ascitic fluid analysis . SBP was defined as polymorphonuclear leucocyte count (PMN) >250/mm3 in ascitic fluid, . Not all cases are associated with positive ascitic fluid cultures.

There are variants of ascitic fluid infections as culture-negative neutrocytic ascites, monomicrobial non-neutrocytic bacterascites, polymicrobial bacterascites and secondary bacterial peritonitis.

The advent of the SBP carries a poor prognosis where the hospital mortality ranged from 10 to 50%. As a consequence, any patient with SBP should be assessed for liver transplantation. Immediate treatment with antibiotics and IV albumin should be initiated.

Studies were conducted on alternatives of the ascitic PMN count as high sensitivity C-reactive protein (hsCRP), serum procalcitonin, urinary lipocalin, ascitic lactoferrin, homocysteine and fecal or ascitic calprotectin.

The gold standard test for SBP is ascitic fluid analysis with measurement of the PMN. It is useful for the diagnosis and monitoring of treatment. The culture of the ascitic fluid may be positive if was done correctly .

There is a variant of SBP that is called culture-negative neutrocytic ascites. It is characterized by elevated ascitic fluid PMN but the culture is negative. It is managed exactly as classic SBP. Such cases would be missed if cultures were not done The manual PMN counting is time consuming, laborious and required some experience to avoid intra- and inter-observer variability. So, a simple rapid bedside test would be useful clinically.

Calprotectin is acute-phase inflammatory protein that is released from the PMN. Calprotectin has anti-proliferative and antimicrobial properties. Calprotectin is used clinically widespread in the diagnosis and monitoring treatment of inflammatory bowel disease .

ELIGIBILITY:
Inclusion Criteria:

-

The patients were divided into two groups:

1. Non-SBP group: it included 25 patients with cirrhotic ascites without clinical or laboratory evidence of SBP.
2. SBP group: it included 25 patients with cirrhotic ascites with SBP. They were diagnosed by positive ascitic fluid bacterial culture, an increase in PMNLs count in ascites (>250 cells/mm3) and without any intra-abdominal source of infection.

Exclusion Criteria:

* (1) Cirrhotic patients with and without SBP receiving antibiotics in last 1 week.

  (2) Recent abdominal surgery (<3 months). (3) abdominal malignancy [hepatocellular carcinoma (HCC), colorectal carcinoma, gastric carcinoma, pancreatic carcinoma, cholangiocarcinoma].

  (4) Intra-abdominal infected lesions, such as abscess, appendicitis, cholecystitis, and pancreatitis.

  (5) History of inflammatory bowel disease (Crohn's disease, ulcerative colitis).

  (6) patients with heart failure (HF), hematological, and autoimmune disorders were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
1-CBC | 6 months
  WBCs count and differential,RBCs count,HB,mcv,Mch,Mchc,platelete count
2-liver function test | 6 months
  AlT,ASt,Albumin,total protein,bilirubin
3-Renal function test | 6 months
  serum create and urea
4-Ascitic fluid analysis(physical,chemical,microscopic) | 6 months
  physical(colour,aspect) chemical(protien,glucose) microscopical(wbcs total and differential,Rbcs),bacterial culture
Ascitic Fluid calprotectin | 6 months
  ascitic fluid calprotectin by ELISA
INR | 6 months
  international normalization time

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Xiol X, Castellvi JM, Guardiola J, Sese E, Castellote J, Perello A, Cervantes X, Iborra MJ. Spontaneous bacterial empyema in cirrhotic patients: a prospective study. Hepatology. 1996 Apr;23(4):719-23. doi: 10.1002/hep.510230410. PMID 8666323
- [Background] Bernardi M. Spontaneous bacterial peritonitis: from pathophysiology to prevention. Intern Emerg Med. 2010 Oct;5 Suppl 1:S37-44. doi: 10.1007/s11739-010-0446-x. PMID 20865473
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Background] Marciano S, Diaz JM, Dirchwolf M, Gadano A. Spontaneous bacterial peritonitis in patients with cirrhosis: incidence, outcomes, and treatment strategies. Hepat Med. 2019 Jan 14;11:13-22. doi: 10.2147/HMER.S164250. eCollection 2019. PMID 30666172